CLINICAL TRIAL: NCT01306136
Title: Pilot Study of Exposure Therapy for the Treatment of Puerto Ricans With Posttraumatic Stress Disorder
Brief Title: Pilot Study of Exposure Therapy for Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Responsible Party: Mildred Vera, University of Puerto Rico, Medical Sciences Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1300209
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic stress disorder; Prolonged exposure; Cognitive behavior therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged Exposure (Experimental)
  Interventions: Behavioral: Prolonged Exposure
- Usual care (Active Comparator)
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Prolonged Exposure — 15 psychotherapy sessions focused on helping clients overcome avoidance behaviors and emotionally process trauma-related memories
  Arms: Prolonged Exposure
Behavioral: Usual care — Per usual care, patients are referred to a mental health provider within the health care setting.
  Arms: Usual care

SUMMARY:
The purpose of this project is to examine the feasibility of a culturally adapted, manual based Prolonged Exposure therapy intervention for the treatment of Spanish-speaking Puerto Ricans with posttraumatic stress disorder

DETAILED DESCRIPTION:
This project seeks to lay the foundation for an effectiveness trial that will lead to the advancement of treatments for PTSD among Spanish-speaking Latinos, particularly Puerto Ricans. This area of research is important in light of the limited treatment options currently available for Spanish-speakers with PTSD and the long-term negative consequences of this condition. Participants in this study are recruited by referral from mental health providers in a general health setting. Patients meeting criteria for enrollment will be randomly assigned to receive either Prolonged Exposure therapy or treatment as usual. Assessments for all participants will be collected at baseline, week 8, and week 16 after randomization.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PTSD
* CAPS score of at least 45
* 18 to 65 years old
* Spanish speaker
* competent to provide informed consent

Exclusion Criteria:

* history of bipolar disease, schizophrenia or psychotic disorder
* alcohol or drug abuse in the past three months
* moderate to severe traumatic brain injury
* applying for or receiving disability benefits
* clinically judged to have a high acute suicide risk
* life-threatening medical condition
* currently receiving psychotherapy for PTSD or changed psychotropic medication within 2 months of randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale | Baseline, week 8, week 16
  The Clinician-Administered PTSD Scale is a semi-structured interview designed to assess posttraumatic stress disorder (PTSD) diagnostic status and symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Puerto Rico, Medical Sciences Campus, San Juan, Puerto Rico